CLINICAL TRIAL: NCT00100477
Title: Study of Topoisomerase Inhibition in the Treatment of Acute Leukemia
Brief Title: Use of Topotecan in Patients With Refractory Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Immunex Corporation (Industry); SmithKline Beecham (Industry); Amgen (Industry)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: CADE-RCD1
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Non-Hodgkin's Lymphoma; Leukemia
Keywords: Multiple Myeloma; Lymphoma; Leukemia; Etoposide; Drug Therapy; Clinical Trials
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia; Multiple Myeloma; Lymphoma | interventions — Topotecan; Mitoxantrone; Etoposide

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Topotecan; Drug: Mitozantrone; Drug: Etoposide

INTERVENTIONS:
Drug: Topotecan
Drug: Mitozantrone
Drug: Etoposide

SUMMARY:
The purpose of this study is to identify the highest tolerated doses in drugs used to treat aggressive leukemia, lymphoma or multiple myeloma not responding to standard chemotherapy treatment. The drugs being used in this study include drugs frequently used in treating such diseases (mitoxantrone and etoposide) as well as a newer drug that has also been shown to be effective (topotecan).

DETAILED DESCRIPTION:
The purpose of this study is to identify the highest tolerated doses in drugs used to treat aggressive leukemia, lymphoma or multiple myeloma not responding to standard chemotherapy treatment. The drugs being used in this study include drugs frequently used in treating such diseases (mitoxantrone and etoposide) as well as a newer drug that has also been shown to be effective (topotecan).

ELIGIBILITY:
Inclusion Criteria:

Patients in the following disease categories will be considered eligible for this study:

* Any acute leukemia beyond an initial attempt to induce a remission or after relapse
* Chronic Myelogenous Leukemia in Blast Phase
* Refractory Multiple Myeloma
* Refractory non-Hodgkin's and Hodgkin's Lymphoma
* Patients must be more than 14 days beyond prior myelotoxic chemotherapy
* Several other eligibility criteria apply.

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1998-08; Primary Completion 2001-01 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mainwaring, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States